CLINICAL TRIAL: NCT05705492
Title: ACTO: A Phase II, Randomized, Placebo-Controlled Study Evaluating Olanzapine in the Management of Cancer Cachexia
Brief Title: Olanzapine for the Management of Cancer Associated Appetite Loss in Patients With Advanced Esophagogastric, Hepatopancreaticobiliary, Colorectal or Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric Roeland, M.D.,FASCO, FAAHPM, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00024724; P30CA069533 (NIH); NCI-2022-10209 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00024724 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2023-01-06; First posted 2023-01-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Advanced Biliary Tract Carcinoma; Advanced Esophageal Carcinoma; Metastatic Esophageal Carcinoma; Locally Advanced Colorectal Carcinoma; Locally Advanced Esophageal Carcinoma; Locally Advanced Gastric Carcinoma; Metastatic Colorectal Carcinoma (mCRC); Advanced Lung Carcinoma; Locally Advanced Hepatocellular Carcinoma
Keywords: cancer; cachexia; weight loss; loss of appetite
MeSH Terms: conditions — Esophageal Neoplasms; Colorectal Neoplasms; Neoplasms; Cachexia; Weight Loss; Anorexia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (olanzapine, optional biospecimen collection) (Experimental): Patients receive a lower (2.5mg) dose of olanzapine orally (PO) nightly for 12 weeks in the absence of unacceptable toxicity. Patients may choose to enroll in an additional 12 weeks of treatment. Patients can choose to undergo computed tomography (CT) scan at baseline and monthly blood sample collections on study.
  Interventions: Drug: Olanzapine; Other: Questionnaire Administration
- Arm II (Experimental): Patients receive a higher dose (5 mg) of olanzapine PO nightly for 12 weeks in the absence of unacceptable toxicity. Patients may choose to enroll in an additional 12 weeks of treatment. Patients undergo an optional baseline CT scan and collections of monthly blood samples on study.
  Interventions: Drug: Olanzapine; Other: Questionnaire Administration
- Arm III (Placebo Comparator): ARM III: Patients receive placebo PO nightly for 12 weeks in the absence of unacceptable toxicity. Patients may choose to enroll in an additional 12 weeks of treatment. Patients undergo CT scan and monthly collection of blood samples on study.
  Interventions: Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Olanzapine — Given PO
  Other Names: LY 170053; Zyprexa; Zyprexa Zydis
  Arms: Arm I (olanzapine, optional biospecimen collection); Arm II
Drug: Placebo Administration — Given PO
  Arms: Arm III
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well olanzapine works in managing cancer cachexia in patients experiencing esophagogastric, hepatopancreaticobiliary, colorectal, or lung cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic) -associated appetite loss while receiving non-curative cancer therapy. Loss of appetite ("anorexia") in the setting of cancer is a key feature of "cachexia," a syndrome associated with loss of weight and muscle as well as weakness and fatigue. Olanzapine is a drug that targets key neurotransmitters (a type of molecule in the central nervous system that transmits messages to the rest of the body) that may stimulate appetite, restore caloric intake, minimize weight loss, and improve quality of life (QOL).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the impact of olanzapine 2.5 mg versus (vs) placebo on the proportion of patients with locally advanced or metastatic EG, HPB, or lung cancers receiving first-line systemic standard-of-care (SOC) therapy with >5% weight gain over 12 weeks. (Part A)

SECONDARY OBJECTIVE:

I. To evaluate the impact of olanzapine 2.5 mg and placebo vs olanzapine 5 mg on the proportion of patients with >5% weight gain over 12 weeks. (Part A) II. To evaluate the impact of olanzapine 2.5 mg vs olanzapine 5 mg vs placebo on additional cancer cachexia-associated endpoints over 12 weeks (anorexia, nutritional status, physical function, patient-reported symptoms, QOL, safety and toxicity, and healthcare utilization) over 12 weeks. (Part A)

OUTLINE:

PART A: Patients are randomized to 1 of 3 arms. All three arms have an optional baseline computed tomography (CT) scan (timed with standard-of-care imaging) at baseline and optional monthly blood sample collections.

ARM I: Patients receive a lower (2.5 mg) dose of olanzapine orally (PO) nightly for 12 weeks in the absence of unacceptable toxicity. Patients may choose to enroll in an additional 12 weeks of treatment (Part B). Patients may choose to participate to undergo CT scan and collection of blood samples on study.

ARM II: Patients receive a higher (5 mg) dose of olanzapine PO nightly for 12 weeks in the absence of unacceptable toxicity. Patients may choose to enroll in an additional 12 weeks of treatment. Patients may choose to participate to undergo CT scan and collection of blood samples on study.

ARM III: Patients receive placebo PO nightly for 12 weeks in the absence of unacceptable toxicity. Patients may choose to enroll in an additional 12 weeks of treatment. Patients may choose to participate to undergo CT scan and collection of blood samples on study.

PART B: All patients receive a lower (2.5mg) dose of olanzapine PO nightly for 12 additional weeks in the absence of unacceptable toxicity. Patients may choose to participate in additional blood sample collections.

After completion of study treatment, patients are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide written informed consent
* Individuals >= 18 years of age
* Histologically confirmed advanced local or metastatic esophogastric, hepatopancreaticobiliary, colorectal, or lung cancer diagnosis within 12 weeks of screening
* Patients with weight loss as defined by international consensus criteria (documented or patient-reported):

  * ≥ 5% weight loss over the past 6 months
  * ≥ 2% weight loss with body mass index (BMI) <20 kg/m^2 or sarcopenia
* Planned or ongoing first-line palliative antineoplastic therapy (cytotoxic chemotherapy, targeted therapy, immunotherapy, combinations) with or without radiation therapy and have not started the second cycle of first-line palliative antineoplastic therapy. Patients may have received adjuvant antineoplastic therapy at least 6 months prior to screening
* Able to ambulate independently with or without assistive devices (e.g., cane, walker)
* In the case of brain metastases, the individual must be asymptomatic or previously treated with a full cycle of therapy with recovery from any acute effects of radiation therapy or surgery before screening. Such individuals must have discontinued corticosteroid treatment and be neurologically stable for at least 4 weeks before screening
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Able and willing to discontinue the use of any drug or over-the-counter (OTC) product that may interact with the study drug (within a period sufficient for wash-out per the principal investigators [PI's] discretion) and thereafter while on the study
* Willingness to comply with restrictions on chest/breastfeeding
* Individuals capable of childbearing and contributing viable sperm must be willing to comply with contraception requirements and not donate ova or sperm while on the study and for 1 month after that
* A negative pregnancy test at baseline (BL) must be obtained for individuals capable of childbearing

Exclusion Criteria:

* Plan for, or history of (within 30 days of enrollment), the use of an antipsychotic drug, including, but not limited to, risperidone, quetiapine, clozapine, phenothiazine, or butyrophenone. This limitation does not include prochlorperazine and other phenothiazines as antiemetic therapy. The use of antipsychotics concurrent with protocol therapy will not be allowed
* Current use of medications or supplements with the goal of enhancing appetite within ≥14 days, including:

  * megestrol acetate
  * cannabinoids (including, but not limited to dronabinol, medical cannabis, over the counter [OTC] cannabinoid products), and/or
  * Corticosteroids (defined as ≥ 5mg of prednisone [or equivalent per day]), except for standard-of-care chemotherapy-induced nausea and vomiting prophylaxis
* Known history of poorly controlled diabetes, defined as fasting morning blood sugars ≥300 mg/dL or recent hemoglobin A1≥ 8. Individuals with diabetes will undergo hemoglobin A1c (HbA1c) blood testing if they do not have HbA1c results 12 weeks prior to enrollment
* Inadequate organ function, which may include, but is not limited to, the following laboratory results within 28 days before signing consent:

  * Total bilirubin ≥5x upper limit of normal (ULN), aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SPGT]) ≥5X ULN (unless the participant has documented Gilbert's syndrome, hepatocellular carcinoma, or hepatic metastases)
  * Primary investigator (PI) discretion will determine continued eligibility after randomization occurs in the event the liver function test results are above the proposed ULN
  * Renal disease requiring dialysis or calculated glomerular filtration rate (GFR) ≤ 30 mL/minute/1.73 m^2 as calculated by the modification of diet in renal disease (MDRD) equation
* Tube feeding or parenteral nutrition at the time of screening
* Any condition that may negatively impact oral absorption of the study drug (including, but not limited to dysphagia, mucositis, gastrectomy, colitis, bowel obstruction, high output ileostomy) or any plan to undergo an intervention that will render such a condition
* Recurrent ascites unresponsive to medical interventions and requires therapeutic paracentesis
* Uncontrolled symptoms at randomization make the individual unsuitable for the study in the judgment of the PI. If uncontrolled symptoms can be effectively palliated for ≥1 week prior, enrollment may be considered at the discretion of the PI
* Uncontrolled infection, including coronavirus disease 2019 (COVID-19), at time of randomization. Individuals with the uncontrolled infection will not be eligible as the symptomology of infection may obscure the outcomes of this study
* Other medical or psychiatric condition, including recent (within 1 year) or active suicidal ideation/behavior or laboratory abnormality, may increase the risk of study participation or, in the PI's judgment, makes the participant inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients exhibiting weight gain greater 5% | Baseline to 12 weeks from baseline
  >5% weight gain comparing olanzapine 2.5mg (Arm I) vs. placebo (Arm III)

SECONDARY OUTCOMES:
Change in Weight | Baseline to 12 weeks from baseline
  >5% weight gain comparing olanzapine 2.5 mg (Arm I) vs. olanzapine 5mg (Arm II)
  >5% weight gain comparing olanzapine 5 mg (Arm II) vs. placebo (Arm III)
Anorexia | At 12 weeks from baseline]
  Patient reported anorexia comparing olanzapine 2.5 mg (Arm 1) vs. olanzapine 5 mg (Arm 2) vs. placebo (Arm 3) Anorexia will be measured using the Functional Assessment of Anorexia-Cachexia Therapy (FAACT), a 12-item subscale of patients' perceptions of appetite (maximum score of 48, higher scores indicate less anorexia). A FAACT score ≤ 37 indicates anorexia.
Appetite | Baseline up to 12 weeks from baseline
  Change in appetite will be measured using the Visual Analog Scale for appetite (VAS), a 10-point scale with a higher score indicating a better appetite. A ≥3-point improvement in appetite at the end of the 12-week placebo-controlled Part A as compared to baseline in each arm will be considered an improvement in appetite.
Nutrition | At baseline and at 4, 8, 12 weeks from baseline
  Nutritional Status will be measured using the Patient- Generated Subjective Assessment Short Form (PG-SGA-SF); scored on a scale of 0-36 with a higher score indicating worse malnutrition.
Physical Function | At baseline and at 4, 8, and12 weeks from baseline
  Eastern Cooperative Oncology Group (ECOG) Performance Status is a clinician's assessment of physical function rated 0 to 5 with a lower score indicating better performance.
Physical Function | At baseline and at 4, 8, and12 weeks from baseline
  Karnofsky Performance Scale (KPS) is a clinician assessed score (0-100) to evaluate physical function and ability to carry out daily activities. A higher score indicates better performance. [Time Frame: At baseline and at 4, 8, 12 weeks from baseline]
Physical Function | At baseline and at 4, 8, and12 weeks from baseline
  Tthe Short Physical Performance Battery (SPPB) is a physical function assessment consisting of 3 timed measures and scored 0 to 12 with a higher score indicating better performance.
Patient Reported Quality of Life | Baseline to 12 weeks from baseline
  Patient reported quality of life will be measured using the Functional Assessment of Cancer Therapy - General (FACT-G,) consisting of four domains (physical, social, emotional, and functional) of well-being with scores ranging from 0 to 108 with higher scores indicating better QOL.
Patient-reported impression of change | At 12 weeks from baseline
  Patient Global Impression of Change (PGI-C) is a 7-point scale depicting a patient's rating of overall improvement in appetite and fatigue with a higher score indicating more improvement .
Patient Reported Symptoms | At 4, 8, and 12 weeks from baseline
  Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) will be used to capture symptoms associated with cancer cachexia and/or its treatment. Each response is scored from 0-4 with a higher score indicating more severity.
Incidence of adverse events | At 4, 8, and 12 weeks from baseline
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.
Proportion of patients with ≥1 unplanned hospitalization | At baseline and at 4, 8, and 12 weeks from baseline
  Calculation and analysis of patients who have 1 or more unplanned hospitalization.
Proportion of patients with ≥1 emergency department visit | At baseline and at 4, 8, and 12 weeks from baseline
  Health care utilization including emergency department visits, hospital admissions.
Proportion of patients with ≥1 unplanned hospitalization | From baseline to 12 weeks
  Number of unplanned hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Eric Roeland, M.D., FAAHPM, FASCO, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States